CLINICAL TRIAL: NCT02464566
Title: 12 Weeks Intensive Lifestyle Intervention Program in Primary Care Obesity Clinic for Obese Adults: Randomized Control Trial, Jeddah 2015
Brief Title: 12 Weeks Intensive Lifestyle Intervention Program in Primary Care Obesity Clinic for Obese Adults: Jeddah 2015
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saudi Commission for Health Specialties, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Riyad Q. Alghamdi, Dr., Saudi Commission for Health Specialties, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaudiCHS
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- L Group (Experimental): Weekly individual session in obesity clinic (15 to 20 min.) for the first 4 weeks then one individual session in obesity clinic (10 to 20 min.) every two weeks (week 5 to week 12).
  Total sessions in 12 weeks: 8 (including the final data collection visit). The components of the program:
  1) Low carbohydrate (aim to achieve spontaneous reduction in calorie intake) 2) increased physical activity; 3) behavioural strategies to facilitate adherence to diet and activity prescriptions.
  Interventions: Behavioral: Intensive lifestyle intervention; Other: Health Education
- C Group (Active Comparator): One session regarding diet restriction and physical activity with printed health education papers.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention
  Arms: L Group
Other: Health Education

SUMMARY:
With low carbohydrate dietary approach for both arms, the investigators will examine the effectiveness of 12-weeks intensive lifestyle intervention program provided in individual sessions in primary health care obesity clinic in Jeddah with aim to achieve 5% reduction of baseline weight for experimental participants in comparison with active comparator group (only one health education session).

DETAILED DESCRIPTION:
The study has two arms:

Active Comparator Arm:

Only health education. One session regarding diet restriction and physical activity with printed health education papers.

Experimental Arm:

Intensive lifestyle intervention Weekly individual session in obesity clinic (15 to 20 min.) for the first 4 weeks then one individual session in obesity clinic (10 to 20 min.) every two weeks (week 5 to week 12).

Total sessions in 12 weeks: 8 (including the final data collection visit).The components of the program: 1) Low carbohydrate (aim to achieve spontaneous reduction in calorie intake) 2) increased physical activity; 3) behavioral strategies to facilitate adherence to diet and activity prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old or older
* Arabic Male or female
* Body mass index in kg/m2 (BMI) ≥30

Exclusion Criteria:

* Had recent weight loss equal or more than 5% of baseline weight
* Currently take weight loss medication or enrolled in another weight loss program
* Undergone or scheduled (within study duration) weight loss surgery
* History of diabetes, thyroid dysfunction or any other endocrine abnormality, gout, coronary heart disease, stroke, malignancy or psychological condition
* Medical condition that limits ability to comply with the program's physical activity recommendations
* Pregnant or lactating women
* If one participant had recruited in the study, his family members who live with him in the same home will be ineligible (to avoid contamination from the ripple effect on weight loss)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Weight Reduction | 1-12 weeks

SECONDARY OUTCOMES:
Waist circumference changes | 1-12 weeks
Hip circumference changes | 1-12 weeks
Systolic and Diastolic Blood pressure changes | 1-12 weeks